CLINICAL TRIAL: NCT03107897
Title: Prehabilitation for Patients Undergoing Transcatheter Aortic Valve Replacement
Acronym: TAVR-Prehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, James Harvey, Principal Investigator, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAVR Prehab
Record Dates: First submitted 2017-03-07; First posted 2017-04-11 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVR; elevated frailty score; Transcatheter Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Comparing individuals who have prehabilitation prior to their TAVR procedure with those that do not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-procedure standard of care (No Intervention): No prehab prior to TAVR.
- Prehab prior to TAVR procedure. (Active Comparator): Individuals participate in prehabilitation prior to TAVR.
  Interventions: Other: Pre-habilitation

INTERVENTIONS:
Other: Pre-habilitation — Eight - Twelve visits to physical therapy prior to their TAVR procedure.
  Arms: Prehab prior to TAVR procedure.

SUMMARY:
In this pilot study, investigators aim to identify patients undergoing TAVR who are at elevated risk for adverse clinical events due to decreased exertional capacity and physical deconditioning. Investigators aim to determine if monitored pre-procedural physical therapy is safe in these patients. Lastly, investigators aim to assess the efficacy of prehabilitation

1. to improve physical functioning by the time of TAVR and to sustain benefit through 30 days post-procedure; and
2. to determine its effect on post-procedural length-of-stay, clinical outcomes, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ambulatory (with or without an assist device)
* Subject has severe aortic stenosis and is felt an appropriate candidate for TAVR by the Heart Team.
* Subject requires 6.0 seconds or longer to complete a 15ft walk test
* Subject must be able to move between sitting and standing without assistance from another person.
* Subject has adequate iliac and femoral arterial anatomy to allow for TAVR via transfemoral access
* Subject is 18 years of age or greater
* Subject is willing to give consent and participate in the study

Exclusion Criteria:

* Subject is incapable of following instructions
* Subject is unable to meet the minimum required physical therapy visits
* Subject has other medical conditions rendering it unsafe, in the opinion of the Principal Investigator and physical therapy staff, to perform a 6 Minute Walk Test or physical therapy conditioning prior to TAVR
* Subject has significant severe un-revascularized epicardial coronary disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2020-08-09 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity - Change in 6 Minute Walk Test (6MWT) | One month post procedure
  Measure: Does prehabilitation improve the subject's functional exercise capacity from first PT assessment to pre-procedure assessment and first PT assessment to one month post-procedure, as measured by the 6MWT?

SECONDARY OUTCOMES:
Mobility - Timed Up and Go Test (TUG) | One month
  Does prehabilitation improve the subject's mobility from first physical therapy assessment to pre-procedure assessment and first PT assessment to one month post-procedure, as measured by the TUG test?
Balance - Four Square Step Test (FSST) | One month
  Does prehabilitation improve the subject's balance from first physical therapy assessment to preprocedure assessment and first PT assessment to one month post-procedure, as measured by the FSST?
Discharge Disposition | 24-48 hours post procedure
  Does prehabilitation make it less likely that a patient will require a higher level of care at discharge than they require prior to admission (for example, arrive from home and discharged to home)?
Length of stay in the ICU | TAVR procedure admission
  Hours total spent in the ICU for TAVR procedure admission
Total hospital length of stay | TAVR procedure admission
  Days total spent in the hospital for TAVR procedure admission
Change in Quality of Life (KCCQ) | One month
  Does the Kansas City Cardiomyopathy Questionnaire score change from the first physical therapy assessment to one month post-procedure?
30 day readmission | 30 days post procedure
  Does the subject have a 30 day re-admission post-procedure?

CONTACTS AND LOCATIONS:
Overall Officials: James Harvey, MD, Principal Investigator — Wellspan York Hospital
Locations (1):
- Wellspan York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data defined in the protocol will be collected during trial participation and entered in a secured Electronic Data Capturing System. All data shared or copied shared will only occur after complete deidentification. Participant data will be made available for Annual Data Safety Management Board (DSMB) committee review. The Study Protocol, Informed Consent Form, and applicable Case Report Forms will be available.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No End Date
Access Criteria: Researchers who provide a methodologically sound proposal.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03107897/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03107897/ICF_001.pdf